CLINICAL TRIAL: NCT06944132
Title: Adjunctive Use of Topical Cyclosporin A Versus Mitomycin C to Prevent Pterygium Recurrence
Brief Title: CsA vs MMC for Preventing Pterygium Recurrence
Acronym: MMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CsA vs MMC for pterygium; Benha University (Other: Al-Azhar University)
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pterygium; Pterygium of the Conjunctiva and Cornea
Keywords: pterygium; Mitimycin C; Cyclosporin A
MeSH Terms: conditions — Pterygium; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (CsA Group) (Active Comparator): Patients received topical cyclosporin A (0.05%) twice daily for three months postoperatively.
  Interventions: Procedure: Excision of the pterygium; Drug: Post-operative application of CsA
- Group B (MMC Group) (Active Comparator): Patients received a single intraoperative application of mitomycin C (0.02%) for two minutes during surgery
  Interventions: Procedure: Excision of the pterygium; Drug: Intra-operative application of MMC

INTERVENTIONS:
Procedure: Excision of the pterygium — The surgical procedure involved excision of the pterygium, including the fibrovascular head and associated conjunctival tissue, followed by bare sclera closure using an autologous conjunctival graft harvested from the superior bulbar conjunctiva. The graft was secured in place using either fibrin glue or 8-0 absorbable sutures. In Group B, 0.02% mitomycin C (MMC) was applied to the bare sclera for two minutes using a soaked sponge, followed by thorough irrigation with balanced salt solution.
Drug: Post-operative application of CsA — Patients received topical cyclosporin A (0.05%) twice daily for three months postoperatively.
  Arms: Group A (CsA Group)
Drug: Intra-operative application of MMC — 0.02% mitomycin C (MMC) was applied to the bare sclera for two minutes using a soaked sponge, followed by thorough irrigation with balanced salt solution.
  Arms: Group B (MMC Group)

SUMMARY:
aimed to compare the efficacy and safety of topical cyclosporin A (CsA) versus mitomycin C (MMC) as adjunctive therapies in preventing pterygium recurrence after surgical excision.

DETAILED DESCRIPTION:
A total of 40 eyes from 40 patients undergoing pterygium surgery were randomized into two groups: Group A received topical cyclosporin A, while Group B was treated with topical mitomycin C. Ocular surface inflammation scores, recurrence rates, patient-reported symptoms, and adverse effects were assessed at baseline and during follow-up at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with primary pterygium extending at least 1 mm onto the cornea.
* No prior history of pterygium surgery in the affected eye.

Exclusion Criteria:

* History of ocular surface diseases such as dry eye or Sjögren's syndrome.
* Active ocular infection.
* Known hypersensitivity to CsA or MMC.
* Systemic conditions requiring immunosuppressive therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
recurrence rate of pterygium | 6 months after surgery
  the recurrence rate of pterygium, defined as fibrovascular regrowth over the cornea of at least 1 mm

SECONDARY OUTCOMES:
Change in parameter OSDI (ocular surface disease index) from 0 to 100 points. | 6 months after surgery
  OSDI (from 0 to 100 points) where patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time" a final score is calculated which ranges from 0 to 100 with scores and based on their OSDI scores, patients can be categorized as having a normal ocular surface (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) ocular surface disease.
Change in clinical parameter Schirmer test (from 0 to 15 mm) | 6 months after surgery
  The Schirmer test score is determined by measuring the length of the strips' moistened area against fluid movement
Change in clinical parameter (TBUT) | 6 months after surgery
  Change in clinical parameter Tear breakup time (TBUT) from less than 5 to more than 10 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Saad, Lecturer, Principal Investigator — Benha University, Ebsar Eye Center
Locations (1):
- Ebsar Eye Center, Cairo, Egypt, Egypt